CLINICAL TRIAL: NCT03933891
Title: Advanced Magnetic Resonance Technics for the Assessment of Liver Function Before and After Transjugular Intrahepatic Portosystemic Shunt
Brief Title: Magnetic Resonance Technics for the Assessment of Liver Function Before and After TIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Associate Professor, West China Hospital
Other Study IDs: TIPS-MRI
Record Dates: First submitted 2018-09-26; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Liver Cirrhosis; Transjugular Intrahepatic Portosystemic Shunt (TIPS); Functional Magnetic Resonance Imaging
Keywords: TIPS; functional MRI; liver corrhosis; portal hypertension; HVPG
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decompensated liver cirrhosis with TIPS
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: TIPS — TIPS: Established distributary channel between the portal vein and hepatic vein via the jugular vein, portal vein blood directly shunts into the systemic circulation to reduce portal vein pressure to effectively prevent bleeding and refractory ascites.

SUMMARY:
Portal hypertension is the end-stage fatal complications of liver cirrhosis. Decompensated cirrhosis patients can pass through transjugular intrahepatic portosystemic shunt to effectively prevent bleeding and refractory ascites. However, the occurrence of hepatic encephalopathy and liver function failure, infection, bleeding again are main lethality postoperative complications after TIPS. The accurate TIPS shunt is necessary to reduce the incidence of complications and improve the patients' survival rate and survival quality. Hepatic venous pressure gradient (HVPG) is standard to evaluate TIPS preoperative and postoperative hemodynamic change and is also the most important the predictors of decompensation and varicose vein bleeding of liver cirrhosis. Whether there is a kind of noninvasive monitoring method can guide TIPS accurate shunt and evaluate the prognosis of patients.

Magnetic resonance imaging (MRI) has a high soft tissue resolution, time and spatial resolution, abdominal MRI can noninvasively, dynamically detect the liver, spleen, portal system functions, the changes of portal system hemodynamics, blood supply of liver tissue, perfusion and liver cell function, etc.

In order to analyze the liver function and survival of liver cirrhosis patients after transjugular intrahepatic portosystemic shunt, advanced magnetic resonance techniques are used before and after transjugular intrahepatic portosystemic shunt. We will combine a variety of advanced magnetic resonance imaging technology, long-term and dynamic monitor TIPS preoperative and postoperative liver function, blood flow, perfusion, the change of tissue elasticity, and analysis the incidence of hepatic encephalopathy, hemorrhage, hepatic failure and survival rate with MRI changes. Finally, we will develop new prediction index, guide TIPS precision shunts, evaluate a variety of the value of imaging technology in the application of patients with TIPS to find the most sensitive technology, and discover the correlation between MRI function parameters with patient's survival. In order to analyze the liver function and survival of liver cirrhosis patients after transjugular intrahepatic portosystemic shunt, advanced magnetic resonance techniques are used to evaluate liver function, blood flow, elasticity, perfusion of before and after transjugular intrahepatic portosystemic shunt.

DETAILED DESCRIPTION:
Portal hypertension is the end-stage fatal complications of liver cirrhosis. Decompensated cirrhosis patients can pass through transjugular intrahepatic portosystemic shunt to effectively prevent bleeding and refractory ascites. However, the occurrence of hepatic encephalopathy and liver function failure, infection, bleeding again are main lethality postoperative complications after TIPS. The accurate TIPS shunt is necessary to reduce the incidence of complications and improve the patients' survival rate and survival quality. Hepatic venous pressure gradient (HVPG) is standard to evaluate TIPS preoperative and postoperative hemodynamic change and is also the most important the predictors of decompensation and varicose vein bleeding of liver cirrhosis. Whether there is a kind of noninvasive monitoring method can guide TIPS accurate shunt and evaluate the prognosis of patients.

Magnetic resonance imaging (MRI) has a high soft tissue resolution, time and spatial resolution, abdominal MRI can noninvasively, dynamically detect the liver, spleen, portal system functions, the changes of portal system hemodynamics, blood supply of liver tissue, perfusion and liver cell function, etc. Magnetic resonance 4D-flow imaging, can accurately measure the portal vein system blood vessels and shunt channels, blood volume, flow velocity parameters of blood flow can be detected. Recent studies have confirmed that the 4D-flow technology can accurately, long-term follow-up monitoring TIPS preoperative, postoperative portal vein blood flow, which have better sensitivity and more accurate than ultrasound to detect blood flow. Magnetic resonance perfusion imaging of the liver can quantitatively obtain liver tissue microcirculation status, monitor portal vein and hepatic artery blood perfusion, the liver perfusion has a significant correlation with Child-Pugh score and degree of liver fibrosis and cirrhosis of the liver. Compared with the traditional magnetic resonance imaging contrast agents, liver specific contrast agents have small renal toxicity, uptake by liver cell specificity, recent studies have found that magnetic resonance imaging with liver cell specificity contrast agents have significantly correlated with the stage of fibrosis of the liver and liver function, and has been used in the clinical staging of liver fibrosis and early detection of hepatocellular carcinoma (HCC). Magnetic resonance elastography (MRE) is a new imaging technology in recent years and a unique image method. As a noninvasive and quantitative method to detect elastic properties of the organ. Plenty of research results showed that in patients with liver cirrhosis, liver and spleen of elasticity have significant correlation with the degree of portal hypertension. So far, a variety of functional imaging methods grade and guide prognosis of patients with cirrhosis, which have been confirmed to have significant clinical value. MRE has been written for the latest diagnosis and treatment of portal hypertension guidelines.

In order to analyze the liver function and survival of liver cirrhosis patients after transjugular intrahepatic portosystemic shunt, advanced magnetic resonance techniques are used before and after transjugular intrahepatic portosystemic shunt. Researchers will combine a variety of advanced magnetic resonance imaging technology, long-term and dynamic monitor TIPS preoperative and postoperative liver function, blood flow, perfusion, the change of tissue elasticity, and analysis the incidence of hepatic encephalopathy, hemorrhage, hepatic failure and survival rate with MRI changes. Finally, Researchers will develop a new predictive index, guide TIPS precision shunts, evaluate a variety of the value of imaging technology in the application of patients with TIPS to find the most sensitive technology, and discover the correlation between MRI function parameters with patient's survival. In order to analyze the liver function and survival of liver cirrhosis patients after transjugular intrahepatic portosystemic shunt, advanced magnetic resonance techniques are used to evaluate liver function, blood flow, elasticity, perfusion of before and after transjugular intrahepatic portosystemic shunt.

Materials and Methods Patients Inclusion criteria: 18-75 years old; liver cirrhosis (diagnosis by imaging, laboratory examination, clinical symptoms and liver biopsy); history of endoscopy confirmed esophageal varicose vein hemorrhage (5 days or longer); the Child-Pugh, B or C less 13; willing to participate in this clinical study, and sign an Informed consent. Exclusion criteria: Child-Pugh ≥12 or MELD ≥18; non-cirrhotic portal hypertension (including regional portal hypertension); total bilirubin over 2 times upper; combined liver cancer or other malignant tumor; infection, uncontrolled sepsis, etc; There are other contraindications to TIPS, EVL and NSBB treatment; heart, lung, kidney and other organs severe disease; women during pregnancy or lactation.

The patients' information Basic information: name, age, gender, work, BMI, rural/urban; Past medical history: the presence of a stool and hemoptysis, ligation hemostasis under gastroscopy history; History of ascites; Hepatic encephalopathy history; Drugs make: diuretics, B-blocker; With or without cardiopulmonary dysfunction history. Cause: alcoholic liver cirrhosis; HBV/HCV related cirrhosis of the liver; AIH, PBC, others. TIPS surgery reason: gastrointestinal bleeding, ascites, other. TIPS postoperative complications: hepatic encephalopathy, ascites, varicose vein bleeding, kidney failure, liver failure. Before and after TIPS, 96 hours, 1 month, 3 months, 6 months and 12 months, then each half year to follow-up until to 5 years. Physical signs and symptoms, Child-Pugh score, MELD score, ammonia and platelet are collected. Before and after TIPS, 96 hours, 6 months and 12 months, multi parameters MRI is performed. MRI scan parameters: 4D-flow sequence: the respiratory gating and cardiac switch control, phase code acquisition of three- space, to obtain parameters of blood flow parameters mapping images. Imaging parameters: imaging volume, 32 × 32 ×24 cm2 to get the isotropic spatial resolution 1.25 mm. TR/TE: 6.4ms/2.2ms, Flip Angle: 16 °. Imaging time is about 12 minutes, depending on the respiratory gating. MRE: simple principle is on the basis of common MRI scans, install a non-magnetic voltage sensor on patients to produce mechanical vibration that transfer into tissues and organs. Particle produce displacement in the direction of propagation of mechanical vibration. The size of the displacement associated with the level of organization elasticity. Imaging parameters are as follows: 3.0 T MR (GE), 12 channels of the surface phased array coil, respiratory gating, single-shot spin echo planar imaging sequence with flow compensation movement encoding gradient, Mechanical wave frequency, 25, 30, 40, 50, and 60 Hz; the spatial resolution: 2 × 2× 2.5 mm3, FOV: 384 x 256; repetition time: 1820 ms; echo time: 54 ms; Matrix: 192 x 128; Perfusion MRI: a 2D fast spoiled gradient echo multi flip-angle T1 map was produced before contrast agent injection with FOV: 60×60×40 mm3; thickness: 2.0 mm; TR：12.4 ms; TE：2.1 ms; matrix: 256 × 128; NEX: 1; with different flip angle 5°, 10°, 20°, 30°, 40°, 50°. The parameters of DCE-MRI were the same as those above, except the flip angle was 30°, after six phase baseline images, 0.025mM/kg Gd of Gd-EOB-DTPA, then 40 phase images were acquired. Liver specificity contrast agents enhanced imaging parameters: 3.0T MR, 12 channels on the surface phased array coil, VIBE: Volume Interpolated Breath-hold Examination, repetition time: 3.1 ms; echo time: 1.16 ms; reconstruction resolution size: 1.3 ×1. 3 × 1.3 mm3; The scanning resolution: 1.7 ×1. 3 ×1. 3 mm3. The MR functions parameters are collected: the liver, the spleen elasticity; 4 D-flow: the superior mesenteric vein (SMV), splenic vein (SV), portal vein (PV) of flow volume, pulse wave velocity (PWV); Perfusion: rCBV, rCBF, MTT; T1 mapping: liver, spleen and kidney T1 values; Magnetic resonance liver cell specificity of contrast agents enhancement: arterial phase, portal phase, liver and gall T1WI signal value of liver tissue. The MR function parameter changes as followed after TIPS will be analyzed. The MR function parameters with chemical biomarkers to predict survival will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old;
* Liver cirrhosis (diagnosis by imaging, laboratory examination, clinical symptoms and liver biopsy);
* History of endoscopy confirmed esophageal varicose vein hemorrhage (5 days or higher);
* The Child-Pugh, B or C less 13;
* Willing to participate in this clinical study, and sign an informed consent.

Exclusion Criteria:

* Child-Pugh ≥12 or MELD ≥18;
* Non-cirrhotic portal hypertension (including regional portal hypertension); total bilirubin over 2 times upper;
* Combined liver cancer or other malignant tumor;
* Infection, uncontrolled sepsis, etc.;
* Heart, lung, kidney and other organs, severe disease;
* Women during pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Decompensated liver cirrhosis, secondary prevention with TIPS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-08-28 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 5 years
Incidence of hepatic encephalopathy | 5 years
Varices rebleeding rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD，PhD, Study Director — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China